CLINICAL TRIAL: NCT07294573
Title: Maternal Health Assessment and Clinical Referral Integrated Into Pediatric Care (M-HARP) in the Dominican Republic
Brief Title: Maternal Health Assessment in Pediatric Care
Acronym: M-HARP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: John James Parker (Other)
Collaborators: Clínica de Familia La Romana, Dominican Republic (Unknown)
Responsible Party: Sponsor-Investigator, John James Parker, Assistant Professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00224392; 1001PC (Other Grant/Funding Number: Northwestern Institute for Global Health)
Record Dates: First submitted 2025-12-08; First posted 2025-12-19 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Postpartum Care; Primary Care; Mental Health; Family Planning; Care Coordination
MeSH Terms: conditions — Psychological Well-Being | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention)
- M-HARP recipient (Experimental): Participants will complete a brief health questionnaire and will be referred to clinical care if indicated.
  Interventions: Behavioral: referral

INTERVENTIONS:
Behavioral: referral — Participants in the intervention arm will be given the "M-HARP questionnaire." The M-HARP questionnaire will gather information on healthcare visits since delivery, desire for contraception, depression screening, and desire for referral. The M-HARP questionnaire will be subsequently reviewed by the pediatrician. If the participants meet the criteria, they will be referred to the appropriate clinical service, including primary care, obstetrics and gynecology, family planning and psychological care.
  Arms: M-HARP recipient

SUMMARY:
The major goal of this study is to develop and pilot M-HARP (Maternal Health Assessment and Referral Integrated into Pediatric Care). M-HARP will adapt a successful US-based health screening and referral protocol to fit the needs of new mothers at Clínica de Familia La Romana, Dominican Republic.

DETAILED DESCRIPTION:
The major goal of this project is to improve the access and utilization of primary healthcare of women in the postpartum period at Clínica de Familia La Romana (CFLR), by designing and piloting M-HARP. Additionally, by applying best practices in implementation science, our study will provide data that can be utilized in other settings. First, the investigators will develop strategies for integrating M-HARP into CFLR through stakeholder engagement. Second, we will pilot M-HARP at CFLR by recruiting postpartum women during their child's pediatric well child visit and measure implementation outcomes guided by the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework.

Aim 1: Develop strategies and processes for establishing M-HARP into CFLR. In Aim 1 the investigators will conduct two in-person advisory meetings, each held at CFLR. One meeting will be with mothers that receive their obstetric care and/or bring their children to CFLR for pediatric care. A second meeting advisory meeting clinicians at CFLR- obstetricians, pediatricians, family planning providers, family medicine and internal medicine. In each meeting we will review the M-HARP questionnaire, the draft protocol and conduct a patient journey mapping exercise. These meetings will be audio recorded and transcribed so the meetings can be reviewed later. Results from these meetings are solely recommendations for M-HARP protocol optimization and will not be published. Therefore, the advisory board members are not research participants.

Aim 2: Pilot M-HARP:

The pilot will enroll participants into two separate groups- the standard of care (SOC) group or M-HARP receipt group. All participants are mothers that will be recruited and enrolled while accompanying their infant to a pediatric visit at CFLR. Potential participants will be recruited after their child has been placed in the clinical exam room. In standard practice, the nurse or medical assistant from CFLR will intake the child (record vital signs and review immunization history). Then the family will wait in the exam room for the pediatrician. At this time the research assistant will approach the mother and assess interest in participating in the study. If the mother is interested, the research assistant will explain the study and assess the mother's eligibility. If mother agrees to participate, consent will be explained and signed. This will all occur in the exam room, which is a private space.

In phase 1, the investigators will enroll SOC, who will complete a questionnaire on demographics and medical history but will not have the M-HARP questionnaire reviewed by the pediatrician. Phase 2 will consist of M-HARP recipient group enrollment. During Phase 2, participants will also fill out a questionnaire on demographics and medical history but will also be given the M-HARP questionnaire. The M-HARP questionnaire will gather information on healthcare visits since delivery, desire for contraception, PHQ-2 depression screening, and desire for referral. The M-HARP questionnaire will be subsequently reviewed by the pediatrician. If the participants meet the criteria, they will be referred to the appropriate primary care service within the CFLR clinic. CFLR provides many different care services including primary care, obstetrics and gynecology, family planning and psychological care. Follow-up for SOCs and M-HARP recipients will occur 2-3 months after enrollment. All participants will be contacted to complete a survey (online or over the phone), which will be a repeat of the M-HARP questionnaire that assesses use of primary care and/or family planning services. At this time, study team members will review Clinical de Familia's medical records to evaluate if participants had scheduled or attended clinical visits. After the follow-up survey, we will conduct interviews with 15 participants in the M-HARP recipient group. The interview will assess the participants' experience in M-HARP, its acceptability, feasibility, and integration into pediatric care at CFLR. Participant information will be de-identified during data analysis and contact information will only be accessible to research staff to ensure confidentiality. Lastly, to ensure that all participants have the same access to health resources, after the follow-up survey the SOC participants will be provided with the same referrals that were offered to the M-HARP recipient group after the initial questionnaire, but their health care use data will not be tracked after that time.

ELIGIBILITY:
Inclusion Criteria:

* Women attending pediatric visits at Clínica de Familia La Romana during the study period
* Women in postpartum period, with children up to 6 months of age ≥18 years

Exclusion Criteria:

* Pregnant with another child, since they will be triaged to prenatal care rather than postpartum primary care
* Unwilling and unable to consent
* Women who do not speak Spanish or Creole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Adoption | From enrollment to one week after enrollment
  Adoption will be measured by the percentage of pediatricians that document review of questionnaire along with the percentage of women that complete the entire questionnaire once enrolled

SECONDARY OUTCOMES:
Effectiveness | from enrollment until 6 months from enrollment
  Effectiveness will be measured by the difference in receipt of postpartum primary care services between in the M-HARP intervention group and the standard of care control group after the study period. Additionally, the proportion of women who are on desired contraceptives between groups is a second effectiveness outcome.
Reach | from enrollment until completion of baseline questionnaire
  Reach will be measured by determining how many women who attend their infants well child visit have already consulted with a primary care service after delivery. This information is collected in the first question of the M-HARP questionnaire.
Implementation | from enrollment to 6 months after enrollment
  Implementation will be measured by determining the number of referrals given if participant met referral criteria. Additionally, if participants subsequently made referral appointment
Maintenance | from enrollment to 6 months following enrollment
  Maintenance will be measured by the number of women who attend primary care appointments after referral. Additionally, it will be assessed by a qualitative discussion with board of key constituents on its maintenance and integration at the clinic after the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica De Familia, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: No